CLINICAL TRIAL: NCT01731457
Title: Limitation of Ischemic Injury of a Kidney Stored in Machine Perfusion in Hypothermia - Evaluation of the Impact on Kidney Allograft Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Piotr Domagała, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N N403 589338-WUM-PD-Poland
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2016-12

CONDITIONS: Transplanted Kidney Ischemia Reperfusion Injury
Keywords: ischemia, reperfusion, kidney, transplantation
MeSH Terms: conditions — Ischemia | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Etanercept (Experimental)
  Interventions: Drug: etanercept
- Control (No Intervention)

INTERVENTIONS:
Drug: etanercept — adding appropriate dose of etanercept to the perfusion fluid
  Arms: Etanercept

SUMMARY:
The aims of this study are:

1. assessment of ischemia injury of kidney retrieved from standard and expanded criteria deceased donor before transplantation
2. assessment of efficacy of kidney ischemia injury decreasing
3. assessment of influence of kidney ischemia injury decreasing on its function after transplantation For the purpose of this research one hundred kidney will be retrieved from deceased donors (standard and expanded criteria deceased donors) for transplantation. All kidneys before transplantation will be stored in machine perfusion in hypothermia with continuous flow - Organ Recovery Systems LifePort - each single kidney in self-contained perfusion system.

For the kidney allograft assessment will be used measurements performed during machine perfusion in hypothermia: renal flow, resistance, lactate dehydrogenase, lactates and ischemia injury markers measured in the fourth hour of perfusion in perfusion fluid.

For kidney ischemia injury assessment such markers will be measured: tumour necrosis factor (TNF alfa), interleukin 2 (IL-2), interleukin 6 (IL-6), high sensitivity C-reactive protein (hsCRP), platelet-derived growth factor (PDGF), cystatin C, kidney Injury Molecule (KIM-1), neutrophil Gelatinase-associated Lipocalin (NGAL), complement component C3, caspase 3.

Every time from pair of retrieved kidneys each kidney will be randomise for one of the group:

* group 1) - 50 kidneys - examined group - "cured" with etanercept (ENBREL) in the first hour of perfusion by adding drug to perfusion fluid,
* group 2) - 50 kidneys - control group - without intervention. Ischemia injury markers will be measured in perfusion fluid by kidney two times (in the first and fourth hour of perfusion) for assessment of efficacy kidney ischemia injury decreasing.

Results of measurements of kidney ischemia injury before transplantation, parameters during machine perfusion in hypothermia and donor parameters will be correlated with kidney allograft function post transplantation.

Immediate, delayed and slow graft function, primary non-function, kidney function assessed by creatinine concentration and creatinine clearance at one day, seven days, two weeks, 1, 6 and 12 months post transplantation and kidney graft survival 6 and 12 months post transplantation will be analysed.

ELIGIBILITY:
Inclusion Criteria:

DONOR STAGE

* donor after brain death
* seronegative HCV (hepatitis C virus)
* procurement of two kidneys from the same donor
* donor center distance up to 220 kilometres from Warsaw
* availability of fluid KPS-1 and cartridge of Organ Recovery System

RECIPIENT STAGE

* recipient of kidneys from deceased donor
* at least eighteen recipient
* expression of informed consent

Exclusion Criteria:

DONOR STAGE

* live kidney donor
* seropositive HCV (hepatitis C virus)
* get only one from the kidneys
* "doubtful" donor - e.g. need for biopsy because of proteinuria or due to histological lesions (e.g. tumor)
* donor center distance above 220 kilometres from Warsaw
* lack of fluid KPS-1 and cartridge of Organ Recovery System

RECIPIENT STAGE

* recipient of kidney form living donor
* minor recipient
* no expression of informed consent
* multiple organ recipient
* recipient "EN BLOC" kidneys or two kidneys
* recipient of kidney from donor under 14 years old
* a need of atypical urinary diversion in kidney recipient
* participation in another study at least in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2011-04; Primary Completion 2014-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
delayed graft function | one week
  a need at least one dialysis during first week after transplantation
12 months graft survival | 12 months
  survival of kidney grafts 12 months after transplantation

SECONDARY OUTCOMES:
acute rejection | 12 months
  biopsy proven acute rejection episodes during the first year after transplantation
kidney ischemia injury assessment | 4 hours
  ischemia injury markers measured two times (in the first and fourth hour of perfusion) in perfusion fluid: tumour necrosis factor (TNF alfa), interleukin 2 (IL-2), interleukin 6 (IL-6), high sensitivity C-reactive protein (hsCRP), platelet-derived growth factor (PDGF), cystatin C, kidney Injury Molecule (KIM-1), neutrophil Gelatinase-associated Lipocalin (NGAL), complement component C3, caspase 3

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Domagala, MD, PhD, Principal Investigator — Medical University of Warsaw
Locations (1):
- Department of General Surgery and Transplantation, Warsaw, Masovian Voivodeship, Poland